# PROTOCOL TITLE:

The Scleroderma Patient-centered Intervention Network - Scleroderma Support group Leader EDucation (SPIN-SSLED) Program Trial

NCT03965780 July 18, 2019

#### PROTOCOL TITLE:

The Scleroderma Patient-centered Intervention Network - Scleroderma Support group Leader EDucation (SPIN-SSLED) Program Trial

#### 1. THE NEED FOR A TRIAL

## 1.1 What is the problem to be addressed?

People with rare diseases face the same challenges as those with more common diseases plus unique challenges, including limited disease education and lack of specialized support options. <sup>1-12</sup> Professionally organized support services for common diseases are often available through the healthcare system, <sup>13,14</sup> but are not typically available in rare diseases. <sup>10,15</sup> As a result, many people with rare diseases look to peer-led support groups for disease-specific education and support. <sup>16-20</sup>

| CONSORT Consolidated Standard of Reporting Trials ICC Intra-class Correlation Coefficient PHQ-8 Patient Health Questionnaire-8 OLBI Oldenburg Burnout Inventory PN-RCT Partially Nested Randomized Controlled Trial RCT Randomized Controlled Trial SSc Systemic Sclerosis SPIN-SSLED SPIN Scleroderma Support group Program SPIN Scleroderma Patient-centered Intervention Network | Table 1: Abbreviations | |
|---|---|---|
| ICC Intra-class Correlation Coefficient PHQ-8 Patient Health Questionnaire-8 OLBI Oldenburg Burnout Inventory PN-RCT Partially Nested Randomized Controlled Trial RCT Randomized Controlled Trial SSc Systemic Sclerosis SPIN-SSLED SPIN Scleroderma Support group Program Leader EDucation Program SPIN Scleroderma Patient-centered Intervention Network | CONSORT | Consolidated Standard of |
| PHQ-8 OLBI Oldenburg Burnout Inventory PN-RCT Partially Nested Randomized Controlled Trial RCT Randomized Controlled Trial SSc Systemic Sclerosis SPIN-SSLED SPIN Scleroderma Support group Program SPIN Scleroderma Patient-centered Intervention Network | | Reporting Trials |
| OLBI Oldenburg Burnout Inventory PN-RCT Partially Nested Randomized Controlled Trial RCT Randomized Controlled Trial SSc Systemic Sclerosis SPIN-SSLED SPIN Scleroderma Support group Program Leader EDucation Program SPIN Scleroderma Patient-centered Intervention Network | ICC | Intra-class Correlation Coefficient |
| PN-RCT Partially Nested Randomized Controlled Trial RCT Randomized Controlled Trial SSc Systemic Sclerosis SPIN-SSLED SPIN Scleroderma Support group Program Leader EDucation Program SPIN Scleroderma Patient-centered Intervention Network | PHQ-8 | Patient Health Questionnaire-8 |
| Controlled Trial RCT Randomized Controlled Trial SSc Systemic Sclerosis SPIN-SSLED SPIN Scleroderma Support group Program Leader EDucation Program SPIN Scleroderma Patient-centered Intervention Network | OLBI | Oldenburg Burnout Inventory |
| RCT Randomized Controlled Trial SSc Systemic Sclerosis SPIN-SSLED SPIN Scleroderma Support group Program Leader EDucation Program SPIN Scleroderma Patient-centered Intervention Network | PN-RCT | Partially Nested Randomized |
| SSc Systemic Sclerosis SPIN-SSLED SPIN Scleroderma Support group Program Leader EDucation Program SPIN Scleroderma Patient-centered Intervention Network | | Controlled Trial |
| SPIN-SSLED SPIN Scleroderma Support group Program Leader EDucation Program SPIN Scleroderma Patient-centered Intervention Network | RCT | Randomized Controlled Trial |
| Program Leader EDucation Program SPIN Scleroderma Patient-centered Intervention Network | SSc | Systemic Sclerosis |
| SPIN Scleroderma Patient-centered<br>Intervention Network | SPIN-SSLED | SPIN Scleroderma Support group |
| Intervention Network | Program | Leader EDucation Program |
| 111011 ( 01111011 1 ( 00 ) ( 0111 | SPIN | Scleroderma Patient-centered |
| CCCI CC | | Intervention Network |
| SSULSS Scieroderma Support Group | SSGLSS | Scleroderma Support Group |
| Leader Self-efficacy Scale | | Leader Self-efficacy Scale |
| VSI Volunteer Satisfaction Index | VSI | Volunteer Satisfaction Index |

Support groups provide important benefits to people with burdensome medical conditions.

people with burdensome medical conditions, based on the principle that people who face similar challenges can empower one another through emotional and practical support. <sup>14,21</sup> Support groups may be held face-to-face or online, led by professionals or peers, and have a structured or an unstructured format. Activities typically involve an educational or information-shar ing component and the exchange of emotional and practical support. <sup>14,18-22</sup>

Systemic sclerosis (SSc), or scleroderma, is a rare, chronic, autoimmune connective tissue disease characterized by abnormal fibrotic processes and excessive collagen production. <sup>23-25</sup> Peer-led support groups play an important role for many people with SSc. 17,26 Currently, there are approximately 275 leaders and co-leaders affiliated with our partners: Scleroderma Canada and Canadian provincial organizations, including Sclérodermie Québec; the Scleroderma Foundation (United States); Scleroderma & Raynaud's UK; Scleroderma Australia and Australian state organizations; and Scleroderma New Zealand; almost all are led by people with SSc. <sup>27-30</sup> Many people with SSc, however, cannot access support groups, and many initiated support groups are not sustained due to challenges that could be addressed via leader training. 18,19 Our partner organizations are committed to improving support group quality and access by providing training to existing support group leaders and to new leaders so that they can start groups in underserved areas and via the Internet. Our Scleroderma Patientcentered Intervention Network (SPIN) team has partnered with patient organization leaders and a team of scleroderma support group leaders to develop the Scleroderma Support group Leader EDucation (SPIN-SSLED) Program. The program is a 3-month group videoconference training program, designed to improve skills and self-efficacy, reduce burden, and reduce emotional distress among support group leaders. Our organizational partners have worked with us to develop the program, and they plan to provide the program to support group leaders post-trial.

SPIN-SSLED Protocol, Version 2 July 18, 2019 We recently completed a feasibility trial of the SPIN-SSLED Program,<sup>31</sup> we are requesting ethical approval to conduct a full-scale trial of the SPIN-SSLED Program.

- **1.2 What are the principal research questions to be addressed?** We will evaluate the effect of the SPIN-SSLED Program on support group leaders' self-efficacy (defined as their perceived ability to carry out actions needed to be successful in support group leadership),<sup>32</sup> burnout, satisfaction with leading a support group, and emotional distress.
- <u>1.2.1. Primary objective:</u> To evaluate the effect of the SPIN-SSLED Program on support group leaders' self-efficacy, measured by the Scleroderma Support Group Leader Self-efficacy Scale (SSGLSS)<sup>33</sup> post-intervention.
- <u>1.2.2. Secondary objectives:</u> To evaluate the program's effects on (1) the SSGLSS<sup>33</sup> at 3 months post-intervention; (2) burnout, measured by the Oldenburg Burnout Inventory (OLBI)<sup>34,35</sup> post-intervention and at 3 months post-intervention; (3) leader satisfaction that leading a group is helping others, measured by the participation efficacy subscale of the Volunteer Satisfaction Index (VSI)<sup>36</sup> post-intervention and at 3 months post-intervention; and (4) emotional distress, measured by the Patient Health Questionnaire-8 (PHQ-8)<sup>37,38</sup> post-intervention. In addition, we will evaluate participant satisfaction among those randomized to the program via the Client Satisfaction Questionnaire-8 (CSQ-8) post-intervention.<sup>39,40</sup>
- **1.3 Why is a trial needed now?** Peer support interventions increase positive health behaviours, self-efficacy for disease management, and mental health. In common diseases, peer support services are often organized through the healthcare system, the but these services are less accessible to people with rare diseases. One reason is that there are major obstacles to evaluating and delivering organized support (e.g., support groups, peer support) for people with rare diseases. We searched PubMed using the names of the approximately 7,000 rare diseases listed in Orphanet's Orphadata but did not find a single trial of an organized support program for patients with any rare disease.

Between 15,000 and 20,000 Canadians are affected by SSc,<sup>47</sup> a rare, chronic, autoimmune connective tissue disease.<sup>23-25</sup> Onset typically occurs between the ages of 30 and 50 years, and approximately 80% of people with SSc are women. Abnormal fibrotic processes that occur in SSc can affect multiple organ systems, including the skin, lungs, gastrointestinal tract, and heart and can cause immune dysfunction and vascular injury.<sup>23-25</sup> Common manifestations include Raynaud's phenomenon,<sup>48</sup> esophageal disease and gastrointestinal symptoms, <sup>49,50</sup> and pulmonary disease.<sup>25</sup> People with SSc commonly experience hand function and mobility limitations, pain, fatigue, sleep problems, pruritus, depression, and body image distress from disfigurement (e.g., skin tightening, pigment changes, hand contractures, telangiectasias).<sup>51-62</sup> Presentation is extremely heterogeneous, and course is highly unpredictable.<sup>23-25</sup>

While many people with SSc rely on support groups in order to learn how to better manage physical and emotional aspects of living with the disease, the majority of SSc patients are not able to access these groups. 17-20,27-30 Currently, there are only a handful of support groups delivered via teleconference or videoconference. 27-30 As such, people with SSc must live close enough to a local group and be able to travel to participate. 18,19 When local groups do exist, they are sometimes disbanded due to the leader's health worsening or to issues related to untrained peer leaders. Some patients prefer not to attend SSc support groups because the group in their area is poorly organized or is overly negative. 18,19 Our research in SSc and research in other diseases, including cancer, has established that leading a support group poses significant challenges and a high level of burden for patient leaders, often resulting in burnout. Peer leaders of illness-based support groups report challenges that include practical

difficulties, such as a lack of resources or poor coordination with medical professionals; difficulties with group leadership tasks, such as managing complex group dynamics or dealing with the worsening health or death of group members; and personal challenges, such as balancing personal and group demands, preventing burnout and stress, and managing one's own health condition while supporting others. <sup>18-20,63-67</sup> These challenges are magnified for peer leaders of rare disease support groups, who also face logistical problems related to small numbers of potential group members, even in urban settings, and limited support from healthcare and patient organizations, which are not as well-resourced as organizations for people with more common diseases, such as cancer, heart disease, or arthritis. <sup>20,46</sup>

By providing key knowledge and skills, the SPIN-SSLED Program could improve the ability of SSc peer support group leaders to lead sustainable, effective support groups; reduce emotional and physical toll on leaders; and encourage new leaders to set up support groups where none exist, locally or via the Internet. The program will be delivered by videoconference because in rare diseases, including SSc, support group leaders are widely dispersed geographically. Videoconferencing has been used successfully to train educators, therapists, other health service providers, and parents of children with behavioural difficulties, for instance. Systematic reviews have found that training healthcare service providers via videoconferencing achieves similar learning outcomes as traditional face-to-face models. Most SSc patients use the Internet. As an example, a 2013 study found that 85% of Dutch SSc patients used the Internet to search for information about SSc. In Canada, SPIN uses Internet-based data collection methods to support an international SSc patient cohort (N > 2000) and is currently testing patient self-management tools delivered via the Internet.

1.3.1 Evidence from systematic reviews: We conducted a systematic review of trials that evaluated the effects of training programs for patient leaders of illness-based support groups on the competency, self-efficacy, burden, and emotional well-being of group leaders. Only one RCT met inclusion criteria. That study evaluated confidence and self-efficacy of cancer support group leaders randomized to either 4-month long high-resource (N = 29; website, discussion forum, 2-day face-to-face training) or low-resource (N = 23; website, discussion forum) interventions. The RCT did not find evidence that the high-resource program was more effective. However, the trial was substantially underpowered, not enough information was provided to determine intervention content or how it was delivered, and the risk of bias was high due to methodological limitations. We updated the systematic review through June 4, 2018, but did not identify any additional trials.

1.3.2. Patient interviews and scleroderma support group survey: Prior to developing the SPIN-SSLED Program, to assess need and inform program development, we sought information on (1) reasons why people with SSc attend or do not attend support groups, (2) the perceived benefits and limitations of participating in support groups, and (3) the training and support needs of SSc support group leaders. To do this, our team, which includes researchers, leaders from our partner patient organizations, and a Support Group Leader Advisory Team of 10 SSc support group leaders, conducted a series of studies. 17-20

We first conducted one-on-one interviews with 30 SSc support group leaders, group members, and non-attenders. Then, we developed and disseminated the Scleroderma Support Group Survey. We generated an initial item pool from our interviews and from surveys done with support groups in more common diseases. We worked with our Advisory Team to edit individual items, delete repetitive items or items less relevant for SSc, and generate new items to reflect content important to SSc that were not reflected in the initial item pool. We disseminated the survey to SSc support group leaders, members, and non-attenders from North America and internationally via (1) postings on SSc organization

websites and other social media venues (e.g., Facebook, Twitter); (2) announcements in SSc patient newsletters; (3) emails to support group leaders and members; and (4) postings in SSc-related chat rooms. Approximately 600 North American patients and 700 SSc patients from other parts of the world completed the survey (approximately 45% non-attenders, 40% group members, and 15% leaders). 17-20

From the interviews and survey,<sup>17-20</sup> we learned that important reasons for attending SSc support groups include giving and receiving emotional and practical support, learning how to manage SSc-related challenges, feeling supported by others with a rare disease, and learning about SSc and SSc research from group members and guest speakers. We learned that many people with SSc do not attend support groups due to factors that include not having access to a local support group, being too ill or disabled to travel, and negative perceptions about support groups (e.g., they are too negative, would not provide useful information). Support group leaders consistently reported difficulty performing tasks necessary to successfully initiate and sustain the groups (e.g., publicizing the group), coping with the emotional demands of leading the group, and managing complex group dynamics. Among support group members, 88% indicated that it was important that groups have trained leaders.

Thus, our research made it clear that there is a need for a well-designed and executed trial of a training program for peer leaders of SSc support groups. We recently completed a feasibility trial<sup>31</sup> that demonstrated that delivering the SPIN-SSLED Program is highly feasible and that it meets the training needs of support group leaders. It also provided preliminary evidence that the program has the potential to improve self-efficacy for carrying out leadership tasks, reduce burden on leaders, and improve emotional distress levels in leaders (see section 2.19 for details of SPIN-SSLED Feasibility Trial).

1.4 How will the results of this trial be used? The preliminary research we have conducted, including our feasibility trial, and the SPIN-SSLED Trial, comprise an *integrated knowledge translation* process, in which researchers and stakeholders work together to define research questions, determine the most appropriate methodology, collect data and interpret findings, and disseminate results (<a href="www.cihr-irsc.gc.ca/e/45321.html#a3">www.cihr-irsc.gc.ca/e/45321.html#a3</a>). Our main patient organization partners, Scleroderma Canada and the Scleroderma Foundation, with whom we have a long history of collaboration, are working with our team to ensure that as many people with SSc as possible have consistent access to effective support group services. We have worked closely with them and with our Support Group Leader Advisory Team to design each stage of preliminary research, the SPIN-SSLED Program, and the SPIN-SSLED feasibility and full-scale trials. Recently, patient organizations from the United Kingdom, Australia, and New Zealand joined our team.

Once tested, SPIN-SSLED will be the only peer support group leader training program that has been evaluated in a well-conducted RCT in any disease. If effective, the SPIN-SSLED Program will be implemented immediately by Scleroderma Canada and all other patient organization partners to train and certify peer support group leaders. These organizations have committed to support ongoing training and to provide logistical and other support to groups with certified leaders. Beyond SSc, the SPIN-SSLED Program will be easily adapted for use in other diseases, and our team is committed to working with organizations outside of SSc to develop capacity to provide training for support group leaders.

1.5 Are there any risks or benefits for participants involved in the trial? The proposed trial intervention is of minimal risk. We do not anticipate any safety concerns with the use of the SPIN-SSLED Program. Participation in the SPIN-SSLED Trial will involve weekly online training sessions, completion of online measures, and participation in a post-program interview. Although it is hypothesized that the SPIN-SSLED Program will improve leaders' self-efficacy for performing leader tasks, reduce burnout, and reduce emotional distress, it cannot be guaranteed that leaders will receive SPIN-SSLED Protocol, Version 2

any benefits from this study. However, information learned from this research may lead to more effective SSc support group leader training, which may in turn benefit those living with SSc in the future or people with other diseases. There will be no financial compensation for leaders who are participating in the SPIN-SSLED Trial.

**1.6 Will participants receive a compensation for their participation in the trial?** No compensation is offered to take part in the SPIN-SSLED Trial.

#### 2. THE PROPOSED TRIAL

**2.1 What is the proposed trial design?** The proposed study will be a pragmatic RCT that tests whether the SPIN-SSLED Program improves support group leader outcomes compared to leaders assigned to a waitlist control. Pragmatic RCTs differ from explanatory or mechanistic trials in that they are intended to test the effectiveness of adding an intervention to routine practice in order to inform practice and policy decisions rather than explain intervention mechanisms.<sup>80-82</sup>

Support group leaders assigned to the SPIN-SSLED Program will be individually randomized and then clustered into training groups. Members of each training group will interact during videoconference training modules. Support group leaders assigned to the waitlist control will not be clustered. They will be randomized individually and will only complete trial measures. A standard cluster RCT design is used when interventions are delivered to groups, rather than individuals, in order to account for dependence between individuals within clusters. <sup>83-85</sup> The SPIN-SSLED Trial will need to account for clustering in the intervention arm, but not the control arm. Thus, we will use a partially nested RCT trial design (PN-RCT). <sup>86-88</sup> The PN-RCT design is a hybrid between a conventional RCT with individual participant randomization and a cluster RCT, in which pre-existing clusters (e.g., primary care practices) are randomized to intervention or control arms. In the PN-RCT design, analyses account for dependence within intervention arm clusters, but treat participants assigned to the control arm individually, as in a conventional RCT. <sup>86-90</sup> Although less common in medical research, PN-RCTs are used extensively in educational and behavioural research. <sup>86</sup>

The reason that we will use a waitlist control group that will receive the program post-trial is that our patient organization partners are invested in providing the training program, regardless of trial outcomes, for reasons of organizational liability and in order to support their support group leader community, the members of which have expressed a strong desire to receive training.

The trial will be registered prior to patient enrollment (clinicaltrials.gov) and will be reported in accordance with standards articulated in the Consolidated Standard of Reporting Trials (CONSORT) statement<sup>91,92</sup> and CONSORT extensions for nonpharmacologic trials,<sup>93</sup> cluster trials,<sup>80</sup> pragmatic trials,<sup>80</sup> and e-health trials.<sup>94</sup>

**2.2** What are the planned trial interventions? The SPIN-SSLED Program uses a problem-based learning approach, which is a learner-centered approach that integrates theory and practice by providing necessary knowledge and skills, presenting complex, real-world problems, and working to identify approaches to solving problems. 95-98 Each module, or learning session, will introduce a topic and provide an overview of key information. In modules that involve managing group or individual interactions, videos that we recorded with members of our Support Group Leader Advisory Team will show SSc support group leaders faced with a problem or situation similar to those that training group participants may encounter in their role as a support group leader. Then, there will be a guided discussion among training group participants about possible approaches and solutions.

The SPIN-SSLED Program includes 13 modules that are delivered via videoconference over the course of the 3-month program in weekly 60- to 90-minute sessions. Module topics include (1) The Leader's Role; (2) Starting a Support Group; (3) Structuring a Support Group Meeting; (4) Scleroderma 101; (5) Successful Support Group Culture; (6) Managing Support Group Dynamics; (7) Loss and Grief: The Support Group Leader; (8) Loss and Grief: Supporting Group Members; (9) Advertising and Recruitment for the Support Group; (10) The Continuity of the Group; (11) Supporting Yourself as a Leader; (12) Remote Support Groups; and (13) Transitions in Support Groups. See Appendix 1 for an overview of module content, Appendix 2 for the training manual, Appendix 3 for the participant manual, and Appendices 4-6 for example module PowerPoint slides.

All English-language SPIN-SSLED training groups will be facilitated by one instructor, and the French-language training groups will be facilitated by a second instructor. In addition to the live modules, SPIN-SSLED Program participants will receive a manual that summarizes didactic material from sessions. Based on our previous experience and consistent with previous trials of videoconference training, 6 support group leaders will be assigned to each training group to maximize effective interaction and participation.<sup>68-71</sup> Training sessions will be delivered using the GoToMeeting® videoconferencing platform, a high-performance platform that has been used successfully in similar applications<sup>72,99,100</sup> and that was used successfully in the SPIN-SSLED Feasibility Trial<sup>31</sup> (see section 2.19). Participants will receive an instruction guide relating to the use of the videoconferencing platform to ensure that everyone can log in successfully (see Appendix 7 for the instruction guide). In addition to the videoconference sessions, participants will have access to the secure, monitored SPIN-SSLED online forum to interact with other participants about program content. (See Appendices 8-10 for forum guidelines and the instruction guide on how to use the chatroom and access session recordings). Participants will also have access to an online resource center containing videos and educational activities that leaders can use during their support group meetings (see Appendix 11 for screenshots of the website).

All SPIN-SSLED sessions will be video-recorded and audited for fidelity to the program manual by two members of the research team. We will use standard methods for evaluating intervention fidelity, <sup>101</sup> including observation of entire sessions for a randomly selected sample of 25% of sessions. Raters will evaluate adherence to each session's goals and content. Consistent with best-practice recommendations for assessing treatment fidelity, <sup>101</sup> this will be done using a checklist based on a standardized format adapted for the specific components of the SPIN-SSLED Program manual.

Participants allocated to the waitlist control will be informed that the SPIN-SSLED Program will be provided to those on the waitlist at the end of the trial. During the trial, they will complete trial measures but will not receive any active intervention as part of the trial.

2.3 What are the proposed practical arrangements for recruitment, consent, and allocation of participants to trial groups? At the initiation of the trial, our partners from Scleroderma Canada and Canadian provincial organizations, including Sclérodermie Québec; the Scleroderma Foundation in the United States; Scleroderma & Raynaud's UK; Scleroderma Australia and Australian state organizations, and Scleroderma New Zealand will contact group leaders to describe the SPIN-SSLED Program and will provide the SPIN team with a list of eligible support group leaders. The description will also contain a link to the public SPIN-SSLED page on SPIN's website (www.spinsclero.com/projects/spin-ssled). This webpage describes the SPIN-SSLED program and presents both written and video testimonials from participants that have participated in the feasibility

trial. Additionally, there is also a video introducing and explaining how the program came to be. (See Appendix 12 for a screenshot of the webpage and links to the webpage videos)

SPIN-SSLED personnel will then send an email invitation with a link to a Qualtrics survey containing the consent form, a demographic questionnaire with information about participants' support group experience (e.g., years of experience or new leader), and questions regarding the days and times when the interested group leaders could attend training sessions. In addition to describing the study, the consent form will explain (1) that some group leaders who enroll in the study will be randomly selected every 3 months to participate in the SPIN-SSLED Program and that some others will be allocated to a waitlist; (2) that participants randomized to participate in the program plus those allocated to the waitlist will complete measures online at the time of randomization post-intervention, and 3 months post-intervention; (3) that, depending on the number of leaders who enroll, it is possible that some group leaders who enroll will not be selected to receive the training nor be asked to complete trial measures as part of the control group; and (4) that, enrolled participants who do not receive the training as part of the trial, either because they are selected for the waitlist or because they are not selected for the training group or the waitlist, will be offered the training post-trial per our agreement with our partner patient organizations. For existing support groups with more than one leader, one co-leader will be specified as the primary participant and any others as secondary; only one leader per support group will be eligible for inclusion in the trial, and the secondary leaders will only be enrolled if the primary leader day and time availabilities do not match those that are able to be provided in the trial. Interested leaders will be provided contact information for SPIN-SSLED trial personnel, who will answer any questions they may have during the consent process and over the course of the trial. At the initiation of the trial, we will send up to 3 emails, one per week, to leaders who do not respond to the initial email or enroll in the trial.

There will be 15 total training groups offered. We will deliver the program to 3 training groups simultaneously. Thus, the intervention will be delivered in 5 "waves" with 3 training groups of 6 participants each per wave, plus 18 participants randomized to the waitlist control per wave. Prior to starting a new wave, we will email participants who have not yet been selected for participation in a prior wave to allow them to update their available days and times. We will then determine characteristics (language, day, time) of the training groups that are needed for the new wave.

Interested leaders who provide consent for participation will be entered into different pools based on their availabilities. For each wave, the random selection of leaders to be allocated to the intervention and waitlist trial arms will be conducted by a third-party centralized randomization service, the Griffith Randomisation Service (<a href="https://www151.griffith.edu.au/">https://www151.griffith.edu.au/</a>). External centralized randomization will ensure that the allocation sequence is concealed and not able to be influenced by study investigators. For each of the 3 new training groups within each wave, SPIN-SSLED personnel will provide the Griffith Randomisation Service with an anonymized list of participants (only ID numbers will be provided) who could participate in the training group based on their day and time availabilities. For each of the 3 groups, the service will randomly select 12 participants from the pool of enrolled group leaders available during the designated day and time for the group and will randomly allocate the 6 to the training group and 6 to the waitlist group using block randomization. To maximize sharing of experiences in groups, we will limit the number of new group leaders without prior experience to 1-2 per training group, depending on the number of new leaders who enroll (to be determined). Thus, the maximum number of new leaders per 12 selected will be either 2 or 4, and randomization will be stratified by new and existing leaders.

- All 12 leaders (training group = 6, waitlist= 6) will receive an email invitation including a clickable link to the online survey platform Qualtrics, where they will be asked to complete the study baseline measures. This email will also communicate participants' assignment to the training program or waitlist control. A second email will be sent to leaders allocated to the training group with the date and time of their first training session, the topic of the first session, the program manual, and information on how to login to the SPIN-SSLED videoconferencing system and online chatroom.
- **2.4 What are the proposed methods for protecting against sources of bias?** A potential concern is that participants will not be blinded to intervention status. In most pragmatic trials of training, education, or behavioural interventions, participants cannot be blinded. This is understood as part of the response to being offered a treatment, similar to what occurs in clinical practice. Ro-82 A second concern relates to the potential for contamination if participants randomized to the SPIN-SSLED Program share learning material with participants in the waitlist control. It is not likely that material would be shared between leaders from different support groups. Nonetheless, to attempt to minimize the influence of possible contamination, we will explain this concern to participants in the training arm of the trial and ask them not to share their material or discuss the training sessions with other group leaders.
- **2.5** What are the planned inclusion/exclusion criteria? There are currently approximately 275 leaders or co-leaders affiliated with our partner patient organizations, not counting potential new group leaders. To be eligible, support group leaders must be on one of our partner organizations' lists of current or potential leaders, must be able to use the Internet to access training sessions, and must be able to complete study questionnaires online. In addition to these requirements, we will only enroll one support group leader per support group. In the case where there are multiple leaders for a single group, the co-leaders must come to a decision together on who they would like to be the primary leader and prioritized for enrolment. The leader(s) designated as secondary will only be enrolled if the primary leader in the group does not have any day and time availabilities that match what is offered as part of the trial. Those that are designated as secondary and who do not undergo training will be placed in a separate waitlist to undergo training post-trial.
- **2.6 What is the proposed duration of treatment period?** The program consists of 13 modules that will be delivered weekly over a 3-month period.
- **2.7** What is the proposed frequency and duration of follow up? Trial outcomes will be assessed at the time of randomization, 3 months later (post-intervention), and 6 months later (3 months post-intervention).
- **2.8** What are the proposed primary and secondary outcome measures? A demographics questionnaire will be administered to all participants (intervention group and waitlist group) before the trial. The demographics questionnaire designed for this study includes basic demographic information, such as gender, age and employment status. The questionnaire also includes disease-related variables, such as years since scleroderma diagnosis and questions relating to participant's leadership role, such as years in role as support group leader or status as a new leader.
- <u>2.8.1. Primary outcome</u>: The primary outcome analysis will compare SSGLSS<sup>33</sup> scores between group leaders allocated to the SPIN-SSLED Program versus the waitlist control post-intervention. The SSGLSS is a 32-item scale designed to assess SSc support group leader confidence to successfully perform leader tasks (e.g., organizational skills), manage group and interpersonal interactions, and balance group leadership and self-care needs. The measure reflects the core educational content of the

SPIN-SSLED Program. It utilizes a 6-point Likert scale ranging from 1 (strongly disagree) to 6 (strongly agree), with higher total scores indicating greater self-efficacy.

We developed the SSGLSS with our Support Group Leader Advisory Team and validated it via our patient surveys (see section 1.3.2). Prior to the development of the SSGLSS, there were no existing measures of support group leader self-efficacy. We validated the SSGLSS<sup>33</sup> in two samples of SSc support group leaders (N = 102, N = 55) and found that it had good internal consistency (Cronbach's alpha 0.96 and 0.95) and hypothesis-consistent convergent validity with a burnout measure, the OLBI.<sup>33,34</sup> In our feasibility trial,<sup>31</sup> SSGLSS pre-post difference was large among participants (standardized mean difference = 1.70; 1.1 point difference per item), suggesting sensitivity to change and further supporting its validity (see section 2.19).

- 2.8.2. Secondary outcomes: Secondary outcomes include the SSGLSS 3 months post-intervention and other outcome measures post-intervention and 3 months post-intervention. Leader burnout will be measured by the OLBI, which has been validated in diverse populations (16 items, 4-point scale from 1 = strongly disagree to 4 = strongly agree). 34,35 Leader satisfaction (participation efficacy) will be measured using a modified version of the participation efficacy subscale of the VSI.<sup>36</sup> The original version of the VSI was validated using a sample of volunteers (N = 327) and was found to be reliable and constructually valid. 36 The participation efficacy subscale asks respondents to indicate their level of satisfaction on 7 items using a 7-point Likert scale from 1 (very dissatisfied) to 7 (very satisfied). Emotional distress will be assessed with the PHQ-8.37,38 The PHQ-8 items measure depressive symptoms over the last 2 weeks on a 4-point scale, ranging from 0 (not at all) to 3 (nearly every day) with higher scores indicating more depressive symptoms. The PHQ-8 performs equivalently to the PHQ-9,<sup>37</sup> which is a valid measure of depressive symptoms in patients with SSc.<sup>38</sup> Participant Satisfaction with the SPIN-SSLED Program will be evaluated with the CSQ-8, 39,40 a standardized measure that is used to assess satisfaction with health services. Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction) with total scores ranging from 8 to 32. The CSQ-8 has been widely validated across a range of client populations.<sup>39</sup>
- <u>2.9 How will the outcome measures be measured at follow up?</u> All outcome measures are self-report. At baseline, post-intervention, and 3 months post-intervention, SPIN-SSLED personnel will email participants with a link to a Qualtrics survey that includes outcome measures. If measures are not completed within a week, a reminder email will be sent, followed by a phone call from trial personnel 10 days from the original email. This is the same method that was used in the SPIN-SSLED Feasibility Trial.
- 2.10 What is the proposed sample size and what is the justification for the assumptions underlying the power calculations? We identified several meta-analyses that have evaluated self-efficacy in terms of knowledge acquisition and confidence in implementing skills acquired in training programs. A 2016 Cochrane review reported a standardized mean difference effect size of 0.87 for 4 educational interventions designed to change knowledge of sickle cell disease among patients and caregivers (standardized mean difference = 1.12 with an outlier study removed). Several other meta-analyses have reported effect sizes of between 0.58 and 0.94. SPIN-SSLED feasibility trial, which only included 10 participants, the pre-post change in self-efficacy for carrying out leadership tasks was 1.70. For an assumed effect size of 0.70, a two-tailed test with  $\alpha = 0.05$ , and an intra-class correlation coefficient (ICC) of 0.05, N = 75 would provide  $\geq$  80% power for self-efficacy for carrying out leader tasks. There was no loss to follow-up in our feasibility trial. Assuming 20% loss to follow-up in the proposed trial, we would need to randomize 94 support group leaders. We believe that this is a

conservative power and sample size estimate. First, based on existing systematic reviews and on results of our feasibility trial, we believe that the true effect size is likely larger than 0.70. Second, in cluster RCTs, ICC values for individual patient outcomes are typically lower than our 0.05 estimate, even when different interveners are involved, and we will use the same trainer across groups in each language. If the true ICC is lower than our 0.05 estimate, this will result in greater power than estimated. Third, there was no loss to follow-up in our feasibility trial, and in our previous completed studies in SSc that required follow-up, loss to follow-up has been 10% or less. 58,111

For the secondary outcomes, burnout and emotional distress, based on published meta-analyses, a standardized mean difference effect size of 0.50 represents a clinically meaningful effect size for improvement that has been achieved in training programs for managers, caregivers of chronically ill patients, and parents of children with difficult behaviour. This is also considered a clinically meaningful effect size for patient-reported health outcomes, including depressive symptoms. For effect size = 0.50, a two-tailed test with  $\alpha$  = 0.05, and an ICC of 0.05, N = 146 would provide  $\geq$  80% power for both self-efficacy and patient-reported health outcomes. Assuming 20% loss to follow-up in the proposed trial, we would need to randomize 182 support group leaders.

Members of our Support Group Leader Advisory Team and our patient organization partners have emphasized the importance of evaluating the trial's planned secondary outcomes. Thus, we will attempt to enroll 180 participants total (15 training groups of 6 participants; 90 participants in waitlist control) in order to have sufficient power to adequately evaluate secondary outcomes.

- **2.11 Will health service research issues be addressed?** Because SSc support group leaders, who are mostly people with SSc, have reported in interviews that leading support groups is burdensome and impacts quality of life, we will measure leader burnout with the OLBI, and emotional distress with the PHQ-8. We will not perform a formal economic evaluation, but we will collect detailed resource utilization data and report this descriptively.
- 2.12 What is the planned recruitment rate? How will the recruitment be organized? Over what time period will recruitment take place? What evidence is there that the planned recruitment rate is achievable? We will recruit 180 eligible leaders who are currently affiliated with our organizational partners (approximately 250, excluding co-leaders; 65%) or who are potential leaders not currently leading a group, which will add to the pool of eligible participants. Our patient organizational partners will contact potential participants. We will identify and recruit potential participants starting one to two months prior to initiation of training groups and will continue throughout the trial. We believe that this is feasible. To obtain 10 participants in the feasibility trial (see section 2.19), our partner organizations provided names of 12 possible participants from their lists, and all 12 agreed to participate (although one person withdrew prior to initiation for medical reasons, and we invited one of two from the waitlist to replace that participant).<sup>31</sup> There appears to be a high-level of enthusiasm in the international SSc community about the program. For instance, we have received 10-20 emails since we launched the feasibility trial from other leaders seeking to participate, even though the program was not advertised. Our patient organization partners will advertise the program to leaders, will emphasize their support, and will explain that the program will enable leaders to be certified, which our organizational partners plan to require for organizational affiliation.
- **2.13** Are there likely to be any problems with compliance? On what evidence are the compliance figures based? Of the 10 participants in the feasibility trial (see section 2.19), 2 participants missed 2 of 13 sessions (hospitalization, vacation), and 3 participants missed 1 session each. Overall, session

attendance was 95% (123 of 130 sessions). All 10 participants completed all baseline and post-trial measures.<sup>31</sup> Thus, we believe that compliance concerns will be minimal.

- **2.14** What is the likely rate of loss to follow up? On what evidence is the loss to follow-up rate based? We believe that the loss to follow-up will be low based on our feasibility trial results (no loss to follow-up) and previous studies in SSc. In a study of depression, for instance, where patients were recruited from multiple centers around Canada and completed burdensome telephone interviews, follow-up one-month post-baseline was completed by 309 of 345 participants (90%). 58,111 We have conservatively estimated a 20% loss to follow-up.
- **2.15 How many centers will be involved?** We will recruit participants from lists provided by Scleroderma Canada and Canadian provincial organizations, including Sclérodermie Québec, the Scleroderma Foundation (United States), Scleroderma & Raynaud's UK, Scleroderma Australia and Australian state organizations, and Scleroderma New Zealand.
- **2.16 What is the proposed type of analyses?** Analyses will be conducted by a statistician blind to trial arm allocation. For the primary outcome analysis (SSGLSS post-intervention), we will use an intent-to-treat analysis that compares all patients randomly allocated to the SPIN-SSLED Program to all patients allocated to the waitlist control. Intervention effect will be estimated using a generalized linear random effects model, adjusted for baseline SSGLSS scores. The model will include a random effect to account for clustering of participants in the training groups, but not for participants in the waitlist control arm. <sup>89,91</sup> We will investigate the effects of missing data using multiple imputation analysis. As a secondary analysis, we will examine SSGLSS scores post-intervention adjusted for baseline participant SSGLSS scores, age, sex, whether or not the leader has SSc, and new versus experienced leader status. Analysis of the SSGLSS at 3 months post-intervention will similarly be done with two analyses.

Analyses of leader burnout and emotional distress outcomes will only include experienced leaders because new leader would not yet experience burnout or emotional distress due to the burden of leading a group. Analyses of these outcomes will similarly be done (1) controlling for baseline scores only and (2) controlling for baseline scores, age, sex, whether or not the leader has SSc, and new versus experienced leader status.

Statistical significance for all analyses will be determined based on two-sided  $\alpha = 0.05$ .

- **2.17 What is the proposed frequency of analyses?** The analyses described above will be performed once, at the end of the trial. No interim analyses are planned.
- **2.18** Are there any planned subgroup analyses? We will evaluate all outcomes after removing any participants who do not have SSc and, for the SSGLSS, after removing participants who are not current group leaders. We anticipate that well over 90% will have SSc and well over 90% will be current group leaders based on information from our organizational partners. In our feasibility trial, 9 of 10 participants were people with SSc and 10 of 10 were group leaders, including one who recently started.<sup>31</sup>
- **2.19** Has any pilot study been carried out using this design? We conducted a feasibility trial of the SPIN-SSLED Program (NCT03508661) that involved delivery of the SPIN-SSLED Program to two training groups of 5 participants each.<sup>31</sup> Scleroderma Canada and the Scleroderma Foundation each provided our team with names of 6 potential participants. All 12 agreed to participate in the program. We enrolled 10 initially, but one was hospitalized before the trial began; therefore, we thus added one participant who had been wait-listed.

Participant attendance was high (95%; 123 of 130 sessions). All 10 participants completed all baseline and post-trial measures, including an individual interview guided by the Patient Education Materials Assessment Tool for Audiovisual Materials (PEMAT). The interview questions addressed topics related to usability, understandability, organization and clarity of the SPIN-SSLED program. We produced user-friendly instructions for GoToMeeting, the online user-forum, and the SPIN data management platform. No sessions were missed or delayed due to technological difficulties, and time for technological support from our team was between 1-2 hours for the entire program.<sup>31</sup>

Pre-training, the mean (standard deviation [SD]) SSGLSS score, the primary outcome for the planned trial, was 124.4 (22.0), which was similar to the scores of our two international samples from the SSGLSS validation study (N = 102, mean [SD] SSGLSS = 122.9 [21.7]; N = 55, mean SSGLSS = 123.9 [19.4]). Post-training, the mean total score increased to 159.2 (17.1). The standardized mean difference effect size was 1.70, which is considered a large effect size. Items are scored on a 1-6 basis, and the average item score increase pre-post training was 1.1 points. For burnout (OLBI) and emotional distress (PHQ-8), the effect size of post-trial score improvement was between 0.38 and 0.45, which is considered a moderate effect size.<sup>31</sup>

Participant satisfaction was very high. Mean post-training score on the CSQ-8 was 30.6 (2.2). On a per item basis, the mean item score was 3.83 (item range 1-4). On the PEMAT interviews, there were relatively minor suggestions for improving the program, and feedback was extremely positive. The overall mean grade given by participants for the SPIN-SSLED Program was 9.4/10, and all 10 participants indicated they would recommend the program to other support group leaders.<sup>31</sup>

## 3. TRIAL

3.1 What are the arrangements for day to day management of the trial? E.g. randomization, data handling, confidentiality, storage and who will be responsible for coordination. The SPIN team, led by Dr. Thombs and located at the Jewish General Hospital, has the primary responsibility for study design and data analysis, maintaining the protocol and implementation of standard operating procedures, conducting recruitment and providing technical support to participants, overseeing trial progress, coordinating study logistics with organizational partners, preparing and distributing regular progress reports, and monitoring progress.

Outcome measures will be completed using the online surveying tool Qualtrics. Once the online survey data is collected, data will be exported to the statistics software program, IBM SPSS. Cleaning of the data will occur within SPSS by members of the study team. All information obtained about the participants during this study will be treated confidentially within the limits of the law. Only the researchers involved in this project will have access to the survey data. To protect the participants' privacy, upon inclusion in the SPIN-SSLED Trial, a unique participant identification number will automatically be assigned to each participant. An encrypted database will be created for the SPIN-SSLED Program, which includes the patient identification number. Only requests authorized by the principal investigator (Dr. Brett Thombs) will be granted access to this encrypted information. The survey is run through Qualtrics, a company whose computer servers are located in the USA. Data security measures in place at Qualtrics are described in the Qualtrics security statement (<a href="http://www.qualtrics.com/security-statement/">http://www.qualtrics.com/security-statement/</a>). Information obtained from the survey and video recordings of the training sessions used to evaluate fidelity to program will be kept for 10 years on encrypted hard drives by the researchers responsible for this study. Access to the data will be limited to the investigators of the study at the Jewish General Hospital.

3.2 What will be the role of each investigator and co-investigator? As principal investigator, Dr. Thombs will oversee trial conduct, data analysis, and knowledge translation activities, and coordinate collaboration between the research team and partners. Dr. Thombs is the Founder and Director of SPIN, which has a long history of successful collaboration with our partners. His expertise in clinical trials and pragmatic trial designs is reflected in his leadership of an international team that has been funded by CIHR to develop a CONSORT extension for trials conducted in cohorts and existing data sources. 119,120 Ms. Maureen Sauvé (Knowledge User) has SSc, is Past-President of Scleroderma Canada and the Scleroderma Society of Ontario, and leads the patient support work of these organizations. Ms. Kerri Connolly (Knowledge User) is Programs and Services Director for the Scleroderma Foundation and responsible for the foundation's patient support programs. Dr. Linda Kwakkenbos, Assistant Professor, Radboud University, is Co-director of SPIN and will work with Dr. Thombs on day-to-day trial management. Dr. Linda Horwood is a SPIN Postdoctoral Fellow who will work with Dr. Thombs and Dr. Kwakkenbos as coordinator of the trial. Dr. Robert Platt is a biostatistician, Professor, and Albert Boehringer I Chair in Pharmacoepidemiology, McGill University. He has extensive experience in the design and analyses of of RCTs, including cluster trials. He designed and will conduct trial analyses. Dr. Vanessa Malcarne is Professor of Psychology, San Diego State University. She has researched psychosocial adjustment and support mechanisms in SSc for over 20 years. Dr. Ghassan El-Baalbaki is Associate Professor of Psychology, Université du Québec à Montréal. He has expertise in peer support in chronic diseases, including SSc, and in training support group leaders. Dr. Sandra Peláez is an investigator with the Lady Davis Institute for Medical Research, Jewish General Hospital. She studies coping and social support in chronic diseases, including SSc. Drs. Malcarne, El-Baalbaki, and Peláez will oversee training groups and monitor training program delivery fidelity. Dr. Marie Hudson is a rheumatologist and Associate Professor, McGill University, who is expert in SSc. She contributed to design of educational materials, and who will oversee their use in the training program. The SPIN-SSLED Support Group Leader Advisory Team consists of SSc patient support group leaders from Canada (Ms. Catherine Fortune, Ms. Geneviève Guillot, Ms. Michelle Richard, Mr. Ken Rozee, Ms. Maureen Sauvé) and the United States (Mr. Stephen Elrod, Ms. Jacqueline Gerena, Ms. Amy Gietzen, Ms. Karen Gottesman, Ms. Nancy Stephens, Ms. Laura Dyas). Members of the Advisory Team were involved in preliminary research and intervention development and preliminary testing and will be involved in patient outreach and collaboration.

3.3 Describe the trial steering committee and if relevant the data safety and monitoring committee. The trial will be overseen by the SPIN Steering Committee (<a href="https://www.spinsclero.com/en/Team?teamID=0d6dd6a6-8bee-62ed-b515-ff0000ce1efe">https://www.spinsclero.com/en/Team?teamID=0d6dd6a6-8bee-62ed-b515-ff0000ce1efe</a>) along with the trial investigators. The Steering Committee will provide scientific direction for the RCT and will meet periodically to assess its progress. It will be responsible for RCT protocol execution, routine monitoring of data quality, and will meet semi-annually to discuss recruitment and retention and to assess that the trial is meeting key milestones consistent with the timeline.

#### REFERENCES

- 1. Kralik D. The quest for ordinariness: transition experienced by midlife women living with chronic illness. J Adv Nurs. 2002 Jul 1;39(2):146-54.
- 2. Karasz A, Ouellette SC, Haworth Continuing Features Submission. Role strain and psychological well-being in women with systemic lupus erythematosus. Women Health. 1995 Dec 17;23(3):41-57.
- 3. Kole A, Faurisson F. The voice of 12,000 patients: experiences and expectations of rare disease patients on diagnosis and care in Europe. EURORDIS-Rare Diseases Eu; 2009 [cited 2019 Mar 24].325p. Available from: http://www.eurordis.org/IMG/pdf/voice 12000 patients/EURORDISCARE FULLBOOKr.pdf.
- 4. European Organisation for Rare Diseases. Rare diseases: understanding this public health priority. 2005. [cited 2019 Mar 24].14p. Available from: https://www.eurordis.org/IMG/pdf/princeps\_document-EN.pdf.
- 5. Cohen JS, Biesecker BB. Quality of life in rare genetic conditions: a systematic review of the literature. Am J Med Genet A. 2010 May;152(5):1136–56.
- 6. Huyard C. What, if anything, is specific about having a rare disorder? Patients' judgements on being ill and being rare. Health Expect. 2009 Dec;12(4):361–70.
- 7. Nettleton S, Watt I, O'Malley L, Duffey P. Understanding the narratives of people who live with medically unexplained illness. Patient Educ Couns. 2005 Feb 1;56(2):205–10.
- 8. Van Walsem MR, Howe EI, Iversen K, Frich JC, Andelic N. Unmet needs for healthcare and social support services in patients with Huntington's disease: a cross-sectional population-based study. Orphanet J Rare Dis. 2015 Dec;10(1):124.
- 9. Anderson M, Elliott EJ, Zurynski YA. Australian families living with a rare disease: experiences of diagnosis, health services use and needs for psychosocial support. Orphanet J Rare Dis. 2013 Feb 11;8(22):1.
- 10. Dwyer AA. Quinton R, Morin D, Pitteloud N. Identifying the unmet health needs of patients with congenital hypogonadotropic hypogonadism using a web-based needs assessment: implications for online interventions and peer-to-peer support. Orphanet J Rare Dis. 2014 Dec;9(1):83.
- 11. Kasparian NA, Rutstein A, Sansom-Daly UM, Mireskandari S, Tyler J, Duffy J, et al. Through the looking glass: an exploratory study of the lived experiences and unmet needs of families affected by Von Hippel–Lindau disease. Eur J Hum Genet. 2015;23(1):34-40.
- 12. Holtzclaw Williams P. Policy framework for rare disease health disparities. Policy Polit Nurs Pract. 2011 May;12(2):114-8.
- 13. Newman S, Steed L, Mulligan K. Self-management interventions for chronic illness. Lancet. 2004 Oct 23;364(94444):1523-37.
- 14. Davison KP, Pennebaker JW, Dickerson SS. Who talks? The social psychology of illness support groups. Am Psychol. 2000 Fe;55(2):205-17.
- 15. Kwakkenbos L, Jewett LR, Baron M, Bartlett SJ, Furst D, Gottesman K, et al. The Scleroderma Patient-centered Intervention Network (SPIN): protocol for a cohort multiple randomised

- controlled trial (cmRCT) design to support trials of psychosocial and rehabilitation interventions in a rare disease context. BMJ Open. 2013 Aug 1;3(8):e003563.
- 16. Reimann A, Bend J, Dembski B. [Patient-centred care in rare diseases. A patient organisations' perspective]. Bundesgesundheitsblatt Gesundheitsforschung Gesundheitsschutz. 2007 Dec;50(12):1484-93.
- 17. Gumuchian ST, Delisle VC, Kwakkenbos L, Pépin M, Carrier ME, Malcarne VL, et al. Reasons for attending support groups and organizational preferences: the European scleroderma support group members survey. Disabil Rehabil. 2017 Dec;19:1-9.
- 18. Delisle VC, Gumuchian ST, Peláez S, Malcarne VL, El-Baalbaki G, Korner A, et al. Reasons for non-participation in scleroderma support groups. Clin Exp Rheumatol. 2016 Sep 1;34(Suppl 100):56-62.
- 19. Gumuchian ST, Delisle VC, Peláez S, Malcarne VL, El-Baalbaki G, Kwakkenbos L, et al. Reasons for not participating in scleroderma patient support groups: a cross-sectional study. Arthritis Care Res. 2018 Feb;70(2):275-83.
- 20. Delisle VC, Gumuchian ST, El-Baalbaki G, Körner A, Malcarne VL, Peláez S, et al. Training and support needs of scleroderma support group facilitators: the North American Scleroderma Support Group Facilitators Survey. Disabil Rehabil. 2018 Apr 25;1-6.
- 21. Aymé S, Kole A, Groft S. Empowerment of patients: lessons from the rare diseases community. Lancet. 2008 Jun 14;371(9629):2048-51.
- 22. Barg FK, Gullatte MM. Cancer support groups: meeting the needs of African Americans with cancer. Semin Oncol Nurs. 2001 Aug 1(3);17:171-8.
- 23. Seibold J. Scleroderma. In: Harris ED, Budd RC, Firestein GS, Genovese MS, Sergent JS, Ruddy S, Sledge CB, editors. Kelly's textbook of rheumatology. 7th ed. Philadelphia: Elsevier; 2005. p. 1279-308.
- 24. Mayes M. Systemic sclerosis: clinical features. In: Klippel JH, Stone JH, Crafford LJ, White PH, editors. Primer on the Rheumatic Diseases. 13th ed. New York: Springer and Arthritis Foundation; 2008 Jan 23. p. 343-50.
- 25. Wigley FM, Hummers LK. Clinical features of systemic sclerosis. In: Hochberg MC, Silman, A.J., Smolen, J.S., Weinblatt ME, Weismann WH, editors. Rheumatology. 3rd ed. Philadelphia: Mosby; 2003. p.1463-80.
- 26. Kwakkenbos L, Delisle VC, Fox RS, Gholizadeh S, Jewett LR, Levis B, et al. Psychosocial aspects of scleroderma. Rheum Dis Clin North Am. 2015 Aug 1;41(3):519-28.
- 27. Scleroderma Canada [Internet]. Canada: Scleroderma Canada. Find a support group. Scleroderma Canada. [cited 2019 Mar 24]; [full page]. Available from: https://web.archive.org/web/20180904003727/www.scleroderma.ca/Support/Find-A-Support-Group.php (web archive). Accessed March 24, 2019.
- 28. Scleroderma Foundation [Internet]. United States: Scleroderma Foundation. Support groups. Scleroderma Foundation. [cited 2019 Mar 24]; [full page]. Available from: www.scleroderma.org/site/PageServer?pagename=patients\_supportgroups#.Vbec7RZvdFw.

- 29. Scleroderma & Raynaud's UK [Internet]. United Kingdom: Scleroderma & Raynaud's UK. Find support. [cited 2019 Mar 24]; [full page]. Available from: www.sruk.co.uk/find-support/.
- 30. Scleroderma Association of New South Wales. [Internet]. New South Wales: Scleroderma Association of New South Wales. Regional support groups. [cited 2019 Mar 24]; [full page]. Available from: www.sclerodermansw.org/regional-support-groups.
- 31. Thombs BD, Dyas L, Pépin M, et al. Scleroderma Patient-centered Intervention Network Scleroderma Supporg group Leader EDucation (SPIN-SSLED) Program: Non-randomised feasibility trial. Submitted for peer review.
- 32. Bandura A. Self-efficacy: the exercise of control. New York, NY: WH Freeman and Company; 1997.
- 33. Pal NE, Gumuchian ST, Delisle VC, Pépin M, Malcarne VL, Carrier ME, et al. Development and preliminary validation of the Scleroderma Support Group Leader Self-efficacy Scale. J Scleroderma Relat Disord. 2018 Feb;3(1):106-11.
- 34. Demerouti E. Burnout: eine Folge Konkreter Arbeitsbedingungen bei Dienstleistungs- und Produktionstätigkeiten [Burnout: A consequence of specific working conditions among human services, and production tasks]. Frankfurt/Main: Peter Lang; 1999.
- 35. Halbesleben JRB, et al. The construct validity of an alternative measure of burnout: investigating the English translation of the Oldenburg Burnout Inventory. Work Stress. 2005 Jul 1;19(3):208-20.
- 36. Galindo-Kuhn R, Guzley RM. The volunteer satisfaction index: Construct definition, measurement, development, and validation. Journal of Social Service Research. 2002 Mar 11;28(1):45-68.
- 37. Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH, et al. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr 1;114(1-3):163-73.
- 38. Milette K, Hudson M, Baron M, Thombs BD, Canadian Scleroderma Research Group. Comparison of the PHQ-9 and CES-D depression scales in systemic sclerosis: internal consistency reliability, convergent validity and clinical correlates. Rheumatology (Oxford). 2010 Jan 25;49(4):789-96.
- 39. Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979 Jan 1;2(3):197-207.
- 40. Kelly PJ, Kyngdon F, Ingram I, Deane FP, Baker Al, Osborne BA. The Client Satisfaction Questionnaire-8: Psychometric properties in a cross-sectional survey of people attending residential substance abuse treatment. Drug Alcohol Rev. 2018 Jan;37(1):79-86.
- 41. Dale JR, Williams SM, Bowyer V. What is the effect of peer support on diabetes outcomes in adults? A systematic review. Diabet Med. 2012 Nov;29(11):1361-77.
- 42. Parry M, Watt-Watson J. Peer support intervention trials for individuals with heart disease: a systematic review. Eur J Cardiovascular Nurs. 2010 Mar;9(1):57-67.

- 43. Webel AR, OkonskyJ, Trompeta J, Holzemer WL. A systematic review of the effectiveness of peer-based interventions on health-related behaviors in adults. Am J Public Health. 2010 Feb;100(2):247-53.
- 44. Pfeiffer PN, Heisler M, Piette JG, Rogers MA, Valenstein M. Efficacy of peer support interventions for depression: a meta-analysis. Gen Hosp Psychiatry. 2011 Jan 1;33(1);29-36.
- 45. Orphadata [Internet]. [updated 2018 Sep 11, cited 2019 Mar 24]. Available from: www.orphadata.org/cgi-bin/inc/product1.inc.php. Accessed March 24, 2019.
- 46. Delisle VC, Gumuchian ST, Rice DB, Levis AW, Kloda LA, Körner A, et al. Perceived benefits and factors that influence the ability to establish and maintain patient support groups in rare diseases: a scoping review. Patient. 2017 Jun 1;10(3):283-93.
- 47. Bernatsky S, Joseph L, Pineau CA, Belisle P, Hudson M, Clarke AE. Scleroderma prevalence: demographic variations in a population-based sample. Arthritis Rheum. 2009 Mar 15;61(13):400-4.
- 48. Merkel PA, Herlyn K, Martin RW, Anderson JJ, Mayes MD, Bell P, et al. Measuring disease activity and functional status in patients with scleroderma and Raynaud's phenomenon. Arthritis Rheum. 2002 Sep;46(9):2410-20.
- 49. Hong BY, Giang R, Mbuagbaw L, Larche M, Thabane L. Factors associated with development of gastrointestinal problems in patients with scleroderma: a systematic review. Syst Rev. 2015 Dec;4(1):188-96.
- 50. Ntoumazios SK, Voulgari PV, Potsis K, Koutis E, Tsifetaki, Assimakopoulos DA. Esophageal involvement in scleroderma: gastroesophageal reflux, the common problem. Semin Arthritis Rheum. 2006 Dec 1;36(3):173-81.
- 51. Thombs BD, van Lankveld W, Bassel M, Baron M, Buzza R, Haslam S, et al. Psychological health and well-being in systemic sclerosis: state of the science and consensus research agenda. Arthritis Care Res. 2010 Aug;62(8):1181-9.
- 52. Haythornthwaite JA, Heinberg LJ, McGuire L. Psychologic factors in scleroderma. Rheum Dis Clin North Am. 2003;29(2):427-39.
- 53. Bassel M, Hudson M, Taillefer SS, Schieir O, Baron M, Thombs BD. Frequency and impact of symptoms experienced by patients with systemic sclerosis: results from a Canadian national survey. Rheumatology. 2011 Dec 11;50(4):762-7.
- 54. Jewett LR, Haythornthwaite JA, Thombs BD. Psychosocial issues and care for patients with systemic sclerosis. In: Varga J, Denton CP, Wigley FM, Allanore Y, Kuwana M, editors. Scleroderma: From Pathogenesis to Comprehensive Management. 2nd ed. Chicago: Springer. 2012. 743 p.
- 55. Jewett LR, Hudson M, Thombs BD. A 38-year-old woman with elevated muscle enzymes, Raynaud's phenomenon and positive anti-topoisomerase I antibody: Is she depressed? In: Silver RM, Denton CP, editors. Case Studies in Systemic Sclerosis. Chicago: Springer. 2011. 355 p.
- 56. Jewett LR, Kwakkenbos L, Carrier M-E, Malcarne VL, Bartlett SJ, Furst DE, et al. Examination of the association of race/ethnicity and sex with appearance concerns: A Scleroderma Patient-

- centered Intervention Network (SPIN) Cohort Study. Clin Exp Rheumatol. 2016 Jun 28;34 (5):92-9.
- 57. Gumuchian ST, Peláez S, Delisle VC, Carrier ME, Jewett LR, El-Baalbaki G, et al. Exploring emotional distress among people living with scleroderma: a focus group study. PLoS One. 2016 Mar 23;11(3):e0152419.
- 58. Thombs BD, Jewett LR, Kwakkenbos L, Hudson M, Baron M, Canadian Scleroderma Research Group. Major depression diagnoses among patients with systemic sclerosis: baseline and one-month follow-up. Arthritis Care Res. 2015 Mar;67(3):411-6.
- 59. Razykov I, Hudson M, Baron M, Thombs BD, Canadian Scleroderma Research Group. Prevalence and clinical correlates of pruritus in patients with systemic sclerosis: an updated analysis of 959 patients. Rheumatology. 2013;52:2056-61.
- 60. Milette K Hudson M, Körner A, et al. Sleep disturbances in systemic sclerosis: evidence for the role of pain, pruritus, and gastrointestinal symptoms. Rheumatology. 2013;52:1715-20.
- 61. Gholizadeh S, Fox RS, Mills SD, Jewett LR, Thombs BD, Malcarne VL. Coping with the disfigurement of scleroderma: facial, skin, and hand changes. In Varga J, Denton CP, Wigley FM, Allanore Y, Kuwana M, editors. Scleroderma: From pathogenesis to comprehensive management, 2nd ed. Chicago: Springer. 2017. 743 p.
- 62. Jewett LR, Kwakkenbos L, Thombs BD. Psychosocial issues and care for patients with systemic sclerosis. In Varga J, Denton CP, Wigley FM, Allanore Y, Kuwana M, editors. Scleroderma: From pathogenesis to comprehensive management, 2nd ed. Chicago: Springer. 2017. 743 p.
- 63. Butow PN, Ussher J, Kirsten L, Hobbs K, Smith K, Wain G, et al. Sustaining leaders of cancer support groups: the role, needs, and difficulties of leaders. Soc Work Health Care. 2006;42(2):39-55.
- 64. Galinsky MJ, Schopler JH. Negative experiences in support groups. Soc Work Health Care. 1994 Oct 20;20(1):77-95.
- 65. Coreil J, Behal R. Man to man prostate cancer support groups. Cancer Pract. 1999 May;7(3):122-9.
- 66. Kirsten L, Butow P, Price M, Hobbs K, Sundquist K. Who helps the leaders? Difficulties experienced by cancer support group leaders. Support Care Cancer. 2006 Jul 1;14(7):770-8.
- 67. Zordan RD, Juraskova I, Butow PN, Jolan A, Kirsten L, Chapman J, et al. Exploring the impact of training on the experience of Australian support group leaders: current practices and implications for research. Health Expect. 2010 Dec;13(4):427-40.
- 68. Hay-Hansson AW, Eldevik S. Training discrete trials teaching skills using videoconference. Res Autism Spect Disord. 2013 Nov 1;7(11):1300-9.
- 69. Seibert DC, Guthrie JT, Adamo G. Improving learning outcomes: integration of standardized patients & telemedicine technology. Nurs Educ Perspect. 2004 Sep 1;25(5):232-7.
- 70. Xavier K, Shepherd L, Goldstein D. Clinical supervision and education via videoconference: a feasibility project. J Telemed Telecare. 2007 Jun 1;13(4):206-9.

- 71. Marziali E, Donahue P. Caring for others: internet video-conferencing group intervention for family caregivers of older adults with neurodegenerative disease. Gerontologist. 2006 Jun 1;46(3):398-403.
- 72. Fisher WW, Luczynski KC, Hood SA, Lesser AD, Machado MA, Piazza CC. Preliminary findings of a randomized clinical trial of a virtual training program for applied behavior analysis technicians. Res Autism Spect Disord. 2014 Sep 1;8(8):1044-54.
- 73. Johnsson G, Lincoln M, Bundy A, Costley D. A systematic review of technology-delivered disability training and support for service providers: implications for rural and remote communities. Rev J Autism Dev Disord. 2016 Dec 1;3(4):387-98.
- 74. Tomlinson J, Shaw T, Munro A, Johnson R, Madden DL, Phillips R, et al. How does tele-learning compare with other forms of education delivery? A systematic review of tele-learning educational outcomes for health professionals. NSW Public Health Bull. 2013 Nov 28;24(2):70-5.
- 75. van der Vaart R, Repping-Wuts H, Drossaert CH, Taal E, Knaapen-Hans HK, van de Laar MA. Needs for online information and support of patients with systemic sclerosis. Arthritis Care Res. 2013 Apr;65(4):594-600.
- 76. Canadian Research Information System [Internet]. [updated 2012 May 14, cited 2019 Mar 24]. Available from: http://webapps.cihr-irsc.gc.ca/funding/detail\_e?pResearchId=7984938&p\_version=CIHR&p\_language=E&p\_session\_id=.
- 77. Canadian Research Information System [Internet]. [updated 2012 May 14, cited 2019 Mar 24]. Available from: http://webapps.cihr-irsc.gc.ca/funding/detail\_e?pResearchId=7994397&p\_version=CIHR&p\_language=E&p\_session\_id=. Accessed March 24, 2019.
- 78. Delisle VC, Gumuchian ST, Kloda LA, Boruff J, El-Baalbaki G, Körner A, et al. The effect of support group peer facilitator training programs on peer-facilitator and support group member outcomes: a systematic review. BMJ Open. 2016 Nov 1;6(11):e013325.
- 79. Turner KA, Rice DB, Carboni-Jiménez A, Boruff J, Thombs BD. The effectiveness of peer facilitator training and support programs to improve facilitator and group outcomes: an updated systematic review. Sys Rev. 2019;8:67.
- 80. Zwarenstein M, Treweek S, Gagnier JJ, Altman DG, Tunis S, Haynes B, et al. Improving the reporting of pragmatic trials: an extension of the CONSORT statement. BMJ. 2008 Nov 11;337:a2390.
- 81. Roland M, Torgerson DJ. Understanding controlled trials: what are pragmatic trials? BMJ. 1998 Jan 24;316(7127):285.
- 82. Torgerson DJ, Torgerson CJ. Designing randomised trials in health, education, and the social sciences: an introduction. Basingstoke, UK: Palgrave Macmillan; 2008. 256 p.
- 83. Campbell MK, Piaggio G, Elbourne DR, Altman DG, CONSORT Group. Consort 2010 statement: extension to cluster randomized controlled trials. BMJ. 2012 Sep 4;345:e5661.

- 84. Puffer S, Torgerson DJ, Watson J. Cluster randomized controlled trials. J Eval Clin Pract. 2005;11(5):479-83.
- 85. Campbell MK, Mollison J, Steen N, Grimshaw J, Eccles M. Analysis of cluster randomized trials in primary care: a practical approach. Fam Pract. 2000 Apr 1;17(2):192-6.
- 86. Lohr S, Schochet PZ, Sanders E. Partially nested randomized controlled trials in educational research: a guide to design and analysis. Washington, DC: National Center for Education Research; 2014 Jul. 179 p.
- 87. Bauer DJ, Sterba SK, Hallfors DD. Evaluating group-based interventions when control participants are ungrouped. Multivar Behav Res. 2008 Jun 20;43(2):210-36.
- 88. Schweig JD, Pane JF. Intention-to-treat analysis in partially nested randomized controlled trials with real-world complexity. Int J of Res Meth Educ. 2016 Jul 2;39(3):268-86.
- 89. Lee KJ, Thompson SG. The use of random effects models to allow for clustering in individually randomized trials. Clin Trials. 2005 Apr;2(2):163-73.
- 90. Roberts C, Roberts SA. Design and analysis of clinical trials with clustering effects due to treatment. Clin Trials. 2005 Apr 2;2(2):152-62.
- 91. Schulz KF, Altman DG, Moher D, CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010;340:c332.
- 92. Moher D, Hopewell S, Schulz KF, Montori V, Gøtzsche PC, Devereaux PJ, et al. CONSORT 2010 Explanation and Elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010;340:c869.
- 93. Boutron I, Moher D, Altman DG, Schulz KF, Ravaud P. Extending the CONSORT statement to randomized trials of nonpharmacologic treatment: explanation and elaboration. Ann Intern Med. 2008 Feb 19;148(4):295-309.
- 94. Eysenbach G, Consort-EHEALTH Group. CONSORT-EHEALTH: improving and standardizing evaluation reports of web-based and mobile health interventions. J Med Internet Res. 2011 Oct;13(4):e126.
- 95. Boud D, Feletti G. The challenge of problem-based learning. 2d ed. London: Kogan Page; 1997. 344 p.
- 96. Duch BJ, Groh SE, Allen DE. The power of problem-based learning. 1st ed. Virginia: Stylus Publishing; 2001. Why problem-based learning? A case study of institutional change in undergraduate education. 2001 p. 3-11.
- 97. Hmelo-Silver CE. Problem-based learning: what and how do students learn? Educ Psychol Rev. 2004 Sep 1;16(3):235-66.
- 98. Torp L, Sage S. Problems as possibilities: problem-based learning for K-16 education. 2nd ed. Virginia: Association for Supervision and Curriculum Development; 2002. 130 p.
- 99. Hommel KA, Gray WN, Hente E, Loreaux K, Ittenbach RF, Maddux M, et al. The Telehealth Enhancement of Adherence to Medication (TEAM) in pediatric IBD trial: design and methodology. Contemp Clin Trials. 2015 Jul 1;43:105-13.

- 100. Williams LK, McCarthy MC, Burke K, Anderson V, Rinehart N. Addressing behavioral impacts of childhood leukemia: a feasibility pilot randomized controlled trial of a group videoconferencing parenting intervention. Eur J Oncol N. 2016 Oct 1;24:61-9.
- 101. Schoenwald SK, Garland AF, Chapman JE, Frazier SL, Sheidow AJ, Southam-Gerow MA. Toward the effective and efficient measurement of implementation fidelity. Adm Policy Ment Health. 2011 Jan 1;38(1):32-43.
- 102. Schulz KF, Grimes DA. Generation of allocation sequences in randomised trials: chance, not choice. Lancet. 2002 Feb 9:359(9305):516-9.
- 103. Asnani MR, Quimby KR, Bennett NR, Francis DK. Interventions for patients and caregivers to improve knowledge of sickle cell disease and recognition of its related complications. Cochrane Database Syst Rev. 2016;10:CD011175.
- 104. Kaminski JW, Valle LA, Filene JH, Boyle CL. A meta-analytic review of components associated with parent training program effectiveness. J Abnorm Child Psychol. 2008 May 1;36(40):567-89.
- 105. Armour TA, Norris SL, Jack L Jr, Zhang X, Fisher L. The effectiveness of family interventions in people with diabetes mellitus: a systematic review. Diabet Med. 2005 Oct;22(10):1295-305.
- 106. Jiang X, Wang J, Lu Y, Jiang H, Li M. Self-efficacy-focused education in persons with diabetes: a systematic review and meta-analysis. Psychol Res Behav Manag. 2019;12:67-79.
- 107. Zhao FF, Suhonen R, Koskinen S, Leino-Kilpi H. Theory-based self-management educational interventions on patients with type 2 diabetes: a systematic review and meta-analysis of randomized controlled trials. J Adv Nurs. 2017 Apr;73(4):812-33.
- 108. Taljaard M, Donner A, Villar J, et al. Intracluster correlation coefficients from the 2005 WHO Global Survey on Maternal and Perinatal Health: implications for implementation research. Paediatr and Perinat Epidemiol. 2008 Mar;22(2):117–25.
- 109. Smeeth L, Ng ES. Intraclass correlation coefficients for cluster randomized trials in primary care: data from the MRC Trial of the assessment and management of older people in the community. Control Clin Trials. 2002 Aug 1;23(4):409-21.
- 110. Hannan PJ, Murray DM, Jabobs DR Jr., McGovern PG. Parameters to aid in the design and analysis of community trials: intraclass correlations from the Minnesota Heart Health Program. Epidemiology. 1994 Jan 1;5:88-95.
- 111. Jewett LR, Razykov I, Hudson M, Baron M, Thombs BD, Canadian Scleroderma Research Group. Prevalence of current, 12-month and lifetime major depressive disorder among patients with systemic sclerosis. Rheumatology. 2013;52(4):669-75.
- 112. Kaminski JW, Valle LA, Filene JH, Boyle CL. A meta-analytic review of components associated with parent training program effectiveness. J Abnorm Clin Psychol. 2008 May 1;36(4);567-89.
- 113. Collins DB, Holton EF III. The effectiveness of managerial leadership development programs: a meta-analysis of studies from 1982 to 2001. Hum Resour Dev Q. 2004 Jun;15(2):217-48.
- 114. Lundahl B, Risser HJ, Lovejoy MC. A meta-analysis of parent training: moderators and follow-up effects. Clin Psychol Rev. 2006 Jan 1;26(1):86-104.

### THOMBS, BRETT – Ethics Proposal: The Scleroderma Support group Leader Education (SPIN-SSLED) Program

- 115. Sörensen S, Pinquart M, Duberstein P. How effective are interventions with caregivers? An updated meta-Analysis. Gerontologist. 2002 Jun 1;42(3):356-72.
- 116. National Institute for Clinical Excellence. Depression: Management of depression in primary and secondary care. London, England: National Institute for Clinical Excellence; 2004. CG23.
- 117. Fournier JC, DeRubeis RJ, Hollon SD, Dimidjian S, Amsterdam JD, Shelton RC. Antidepressant drug effects and depression severity: a patient-level meta-analysis. JAMA. 2010 Jan 6;303(1):47-53.
- 118. Kirsch I, Deacon BJ, Huedo-Medina TB, Scoboria A, Moore TJ, Johnson BT. Initial severity and antidepressant benefits: a meta-analysis of data submitted to the Food and Drug Administration. PLoS Med. 2008 Feb 26;5(2):e45.
- 119. Kwakkenbos L, Juszczak E, Hemkens LG, Sampson M, Fröbert O, Relton C. Protocol for the development of a CONSORT extension for RCTs using cohorts and routinely collected health data. Res Integr Peer Rev. Accepted for publication.
- 120. Kwakkenbos L, Imran M, McCord KA, Sampson M, Fröbert O, Gale C, et al. Protocol for a scoping review to support development of a CONSORT extension for RCTs using cohorts and routinely collected health data. BMJ Open. 2018 Aug 1;8(8):e025266.